CLINICAL TRIAL: NCT02079922
Title: A Phase 1, Randomized, Double-Blind, Placebo-Controlled Study To Assess The Safety, Tolerability, And Pharmacokinetics Of PF-06678552 After Administration Of Multiple Escalating Oral Doses In Healthy Adult Subjects
Brief Title: A Multiple Dose Study Of PF-06678552 In Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: B7611002
Record Dates: First submitted 2014-03-04; First posted 2014-03-06 (Estimated); Last update posted 2014-07-31 (Estimated); Status verified 2014-07

CONDITIONS: Healthy
Keywords: Multiple Ascending Dose; healthy subjects; Hypercholesterolemia; Hyperlipidemias; Dyslipidemias; Lipid Metabolism Disorders; Metabolic Diseases
MeSH Terms: conditions — Hypercholesterolemia; Hyperlipidemias; Dyslipidemias; Lipid Metabolism Disorders; Metabolic Diseases

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (6):
- Cohort 1 (Experimental): Single dose level of PF-06678552 or placebo every 12 hours (Q12H) for 14 days to investigate the safety, tolerability, and pharmacokinetics.
  Interventions: Drug: PF-06678552; Drug: Placebo
- Cohort 2 (Experimental): Single dose level of PF-06678552 or placebo every 12 hours (Q12H) for 14 days to investigate the safety, tolerability, and pharmacokinetics.
  Interventions: Drug: PF-06678552; Drug: Placebo
- Cohort 3 (Experimental): Single dose level of PF-06678552 or placebo every 12 hours (Q12H) for 14 days to investigate the safety, tolerability, and pharmacokinetics.
  Interventions: Drug: PF-06678552; Drug: Placebo
- Cohort 4 (Experimental): Single dose level of PF-06678552 or placebo every 12 hours (Q12H) for 14 days to investigate the safety, tolerability, and pharmacokinetics.
  Interventions: Drug: PF-06678552; Drug: Placebo
- Cohort 5 (Experimental): Single dose level of PF-06678552 or placebo will be provided either once daily (QD), every 12 hours (Q12H), or every 8 hours (Q8H) for 14 days to investigate the safety, tolerability, and pharmacokinetics.
  Interventions: Drug: PF-06678552; Drug: Placebo
- Cohort 6 (Experimental): Single dose level of PF-06678552 or placebo will be provided either once daily (QD), every 12 hours (Q12H), or every 8 hours (Q8H) for 14 days to investigate the safety, tolerability, and pharmacokinetics.
  Interventions: Drug: PF-06678552; Drug: Placebo

INTERVENTIONS:
Drug: PF-06678552 — PF-06678552 or placebo will be administered as an extemporaneously prepared solution every 12 hours for 14 days.
  Arms: Cohort 1
Drug: Placebo — PF-06678552 or placebo will be administered as an extemporaneously prepared solution every 12 hours for 14 days.
  Arms: Cohort 1
Drug: PF-06678552 — PF-06678552 or placebo will be administered as an extemporaneously prepared solution every 12 hours for 14 days.
  Arms: Cohort 2
Drug: Placebo — PF-06678552 or placebo will be administered as an extemporaneously prepared solution every 12 hours for 14 days.
  Arms: Cohort 2
Drug: PF-06678552 — PF-06678552 or placebo will be administered as an extemporaneously prepared solution every 12 hours for 14 days.
  Arms: Cohort 3
Drug: Placebo — PF-06678552 or placebo will be administered as an extemporaneously prepared solution every 12 hours for 14 days.
  Arms: Cohort 3
Drug: PF-06678552 — PF-06678552 or placebo will be administered as an extemporaneously prepared solution every 12 hours for 14 days.
  Arms: Cohort 4
Drug: Placebo — PF-06678552 or placebo will be administered as an extemporaneously prepared solution every 12 hours for 14 days.
  Arms: Cohort 4
Drug: PF-06678552 — PF-06678552 or placebo will be administered as an extemporaneously prepared solution either once daily (QD), every 12 hours (Q12H), or every 8 hours (Q8H) for 14 days.
  Arms: Cohort 5
Drug: Placebo — PF-06678552 or placebo will be administered as an extemporaneously prepared solution either once daily (QD), every 12 hours (Q12H), or every 8 hours (Q8H) for 14 days.
  Arms: Cohort 5
Drug: PF-06678552 — PF-06678552 or placebo will be administered as an extemporaneously prepared solution either once daily (QD), every 12 hours (Q12H), or every 8 hours (Q8H) for 14 days.
  Arms: Cohort 6
Drug: Placebo — PF-06678552 or placebo will be administered as an extemporaneously prepared solution either once daily (QD), every 12 hours (Q12H), or every 8 hours (Q8H) for 14 days.
  Arms: Cohort 6

SUMMARY:
PF-06678552 is a new compound proposed for the treatment of hypercholesteremia. The primary purpose of this study is to evaluate the safety and tolerability, pharmacokinetics, and pharmacodynamics of multiple oral doses of PF-06678552 in healthy subjects.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male and/or female subjects of non-childbearing potential.
* Body Mass Index (BMI) of 18 to 30.5 kg/m2; and a total body weight >50 kg
* Low density lipoprotein cholesterol between 115 mg/dL and 190 mg/dL

Exclusion Criteria:

* Evidence or history of clinically significant hematological, renal, endocrine, pulmonary, gastrointestinal, cardiovascular, hepatic, psychiatric, neurologic, or allergic disease (including drug allergies, but excluding untreated, asymptomatic, seasonal allergies at time of dosing)

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 38 (Actual)
Dates: Start 2014-03; Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
Assessment of adverse events (AEs), clinical laboratory tests, vital signs (including blood pressure and pulse rate), and cardiac conduction intervals as assessed by 12 lead ECG. | 0 to 24 days post dose

SECONDARY OUTCOMES:
Area Under the Curve From Time Zero to Last Quantifiable Concentration (AUClast) for PF-06644927 on day 1 | 0, 0.25, 0.5, 1, 2, 3, 4, 8, 12 hours post dose
Area Under the Curve From Time Zero to Last Quantifiable Concentration (AUClast) for PF-06644927 on day 7 | 0, 0.25, 0.5, 1, 2, 3, 4, 8, 12 hours post dose
Area Under the Curve From Time Zero to Last Quantifiable Concentration (AUClast) for PF-06644927 on day 14 | 0, 0.25, 0.5, 1, 2, 3, 4, 8, 12 hours post dose
Area Under the Curve during the dosing interval (AUCtau) for PF-06644927 on day 1 | 0, 0.25, 0.5, 1, 2, 3, 4, 8, 12 hours post dose
Area Under the Curve during the dosing interval (AUCtau) for PF-06644927 on day 7 | 0, 0.25, 0.5, 1, 2, 3, 4, 8, 12 hours post dose
Area Under the Curve during the dosing interval (AUCtau) for PF-06644927 on day 14 | 0, 0.25, 0.5, 1, 2, 3, 4, 8, 12 hours post dose
Maximum Observed Plasma Concentration (Cmax) for PF-06644927 on day 1 | 0, 0.25, 0.5, 1, 2, 3, 4, 8, 12 hours post dose
Maximum Observed Plasma Concentration (Cmax) for PF-06644927 on day 7 | 0, 0.25, 0.5, 1, 2, 3, 4, 8, 12 hours post dose
Maximum Observed Plasma Concentration (Cmax) for PF-06644927 on day 14 | 0, 0.25, 0.5, 1, 2, 3, 4, 8, 12 hours post dose
Time to Reach Maximum Observed Plasma Concentration (Tmax) for PF-06644927 on day 1 | 0, 0.25, 0.5, 1, 2, 3, 4, 8, 12 hours post dose
Time to Reach Maximum Observed Plasma Concentration (Tmax) for PF-06644927 on day 7 | 0, 0.25, 0.5, 1, 2, 3, 4, 8, 12 hours post dose
Time to Reach Maximum Observed Plasma Concentration (Tmax) for PF-06644927 on day 14 | 0, 0.25, 0.5, 1, 2, 3, 4, 8, 12 hours post dose
Plasma Decay Half-Life (t1/2) for PF-06644927 on day 14 | 0, 0.25, 0.5, 1, 2, 3, 4, 8, 12, 16, 24, 48 hours post dose
Accumulation ratio for Maximum Observed Plasma Concentration (Rac(Cmax)) for PF-06644927 on day 7 relative to day 1 | 0, 0.25, 0.5, 1, 2, 3, 4, 8, 12 hours post dose
Accumulation ratio for Maximum Observed Plasma Concentration (Rac(Cmax)) for PF-06644927 on day 14 relative to day 1 | 0, 0.25, 0.5, 1, 2, 3, 4, 8, 12 hours post dose
Accumulation ratio for Area Under the Curve during the dosing interval (Rac(AUC)) for PF-06644927 on day 7 relative to day 1 | 0, 0.25, 0.5, 1, 2, 3, 4, 8, 12 hours post dose
Accumulation ratio for Area Under the Curve during the dosing interval (Rac(AUC)) for PF-06644927 on day 14 relative to day 1 | 0, 0.25, 0.5, 1, 2, 3, 4, 8, 12 hours post dose
Amount of PF-06644927 excreted in urine (Ae) on day 14 | 0-12 hours post dose
Percent of dose excreted in urine as PF-06644927 (Ae%) on day 14 | 0-12 hours post dose
Renal clearance of PF-06644927 (CLr) on day 14 | 0-12 hours post dose
Area Under the Curve From Time Zero to Last Quantifiable Concentration (AUClast) for PF-06678552 on day 1 | 0, 0.25, 0.5, 1, 2, 3, 4, 8, 12 hours post dose
Area Under the Curve From Time Zero to Last Quantifiable Concentration (AUClast) for PF-06678552 on day 7 | 0, 0.25, 0.5, 1, 2, 3, 4, 8, 12 hours post dose
Area Under the Curve From Time Zero to Last Quantifiable Concentration (AUClast) for PF-06678552 on day 14 | 0, 0.25, 0.5, 1, 2, 3, 4, 8, 12 hours post dose
Area Under the Curve during the dosing interval (AUCtau) for PF-06678552 on day 1 | 0, 0.25, 0.5, 1, 2, 3, 4, 8, 12 hours post dose
Area Under the Curve during the dosing interval (AUCtau) for PF-06678552 on day 7 | 0, 0.25, 0.5, 1, 2, 3, 4, 8, 12 hours post dose
Area Under the Curve during the dosing interval (AUCtau) for PF-06678552 on day 14 | 0, 0.25, 0.5, 1, 2, 3, 4, 8, 12 hours post dose
Maximum Observed Plasma Concentration (Cmax) for PF-06678552 on day 1 | 0, 0.25, 0.5, 1, 2, 3, 4, 8, 12 hours post dose
Maximum Observed Plasma Concentration (Cmax) for PF-06678552 on day 7 | 0, 0.25, 0.5, 1, 2, 3, 4, 8, 12 hours post dose
Maximum Observed Plasma Concentration (Cmax) for PF-06678552 on day 14 | 0, 0.25, 0.5, 1, 2, 3, 4, 8, 12 hours post dose
Time to Reach Maximum Observed Plasma Concentration (Tmax) for PF-06678552 on day 1 | 0, 0.25, 0.5, 1, 2, 3, 4, 8, 12 hours post dose
Time to Reach Maximum Observed Plasma Concentration (Tmax) for PF-06678552 on day 7 | 0, 0.25, 0.5, 1, 2, 3, 4, 8, 12 hours post dose
Plasma Decay Half-Life (t1/2) for PF-06678552 on day 14 | 0, 0.25, 0.5, 1, 2, 3, 4, 8, 12, 16, 24, 48 hours post dose
Accumulation ratio for Maximum Observed Plasma Concentration (Rac(Cmax)) for PF-06678552 on day 7 relative to day 1 | 0, 0.25, 0.5, 1, 2, 3, 4, 8, 12 hours post dose
Accumulation ratio for Maximum Observed Plasma Concentration (Rac(Cmax)) for PF-06678552 on day 14 relative to day 1 | 0, 0.25, 0.5, 1, 2, 3, 4, 8, 12 hours post dose
Accumulation ratio for Area Under the Curve during the dosing interval (Rac(AUC)) for PF-06678552 on day 7 relative to day 1 | 0, 0.25, 0.5, 1, 2, 3, 4, 8, 12 hours post dose
Accumulation ratio for Area Under the Curve during the dosing interval (Rac(AUC)) for PF-06678552 on day 14 relative to day 1 | 0, 0.25, 0.5, 1, 2, 3, 4, 8, 12 hours post dose
Apparent Oral Clearance (CL/F) of PF-06678552 on day 7 | 0, 0.25, 0.5, 1, 2, 3, 4, 8, 12 hours post dose
  Clearance of a drug is a measure of the rate at which a drug is metabolized or eliminated by normal biological processes. Clearance obtained after oral dose (apparent oral clearance) is influenced by the fraction of the dose absorbed. Clearance was estimated from population pharmacokinetic (PK) modeling. Drug clearance is a quantitative measure of the rate at which a drug substance is removed from the blood.
Apparent Oral Clearance (CL/F) of PF-06678552 on day 14 | 0, 0.25, 0.5, 1, 2, 3, 4, 8, 12 hours post dose
  Clearance of a drug is a measure of the rate at which a drug is metabolized or eliminated by normal biological processes. Clearance obtained after oral dose (apparent oral clearance) is influenced by the fraction of the dose absorbed. Clearance was estimated from population pharmacokinetic (PK) modeling. Drug clearance is a quantitative measure of the rate at which a drug substance is removed from the blood.
Apparent Volume of Distribution (Vz/F) of PF-06678552 on day 7 | 0, 0.25, 0.5, 1, 2, 3, 4, 8, 12 hours post dose
  Volume of distribution is defined as the theoretical volume in which the total amount of drug would need to be uniformly distributed to produce the desired plasma concentration of a drug. Apparent volume of distribution after oral dose (Vz/F) is influenced by the fraction absorbed.
Apparent Volume of Distribution (Vz/F) of PF-06678552 on day 14 | 0, 0.25, 0.5, 1, 2, 3, 4, 8, 12 hours post dose
  Volume of distribution is defined as the theoretical volume in which the total amount of drug would need to be uniformly distributed to produce the desired plasma concentration of a drug. Apparent volume of distribution after oral dose (Vz/F) is influenced by the fraction absorbed.

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer Investigational Site, Brussels, Belgium

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=B7611002&StudyName=A%20Multiple%20Dose%20Study%20Of%20PF-06678552%20In%20Healthy%20Subjects